CLINICAL TRIAL: NCT01176201
Title: An Open-Label Study to Determine ADME of 14C Labeled SLV337 After a Single Dose of an Oral Suspension
Brief Title: 14-C ADME (Absorption, Disposition, Metabolism and Excretion) Study in Man
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abbott Products (Industry)
Responsible Party: Sponsor
Organization: Abbott (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: S337.1.005; 2010-020006-15 (EudraCT Number)
Record Dates: First submitted 2010-07-20; First posted 2010-08-05 (Estimated); Last update posted 2011-08-26 (Estimated); Status verified 2011-08

CONDITIONS: Healthy Subjects
Keywords: SLV337; Diabetes; Relative bioavailability; ADME
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): 400 mg suspension
  Interventions: Drug: SLV337 suspension
- B (Active Comparator): 5 x 200 mg immediate release capsule
  Interventions: Drug: SLV337 capsule

INTERVENTIONS:
Drug: SLV337 suspension — 400 mg experimental
  Arms: A
Drug: SLV337 capsule — 5 x 200 mg immediate release capsule
  Arms: B

SUMMARY:
This is an open-label study to determine the ADME (Absorption, Disposition, Metabolism and Excretion) of 14C labeled SLV337 after a single dose of an oral suspension.

DETAILED DESCRIPTION:
The Absorption, Disposition, Metabolism and Excretion of SLV337 will be investigated after a single dose of an oral suspension of 14C-SLV337.

ELIGIBILITY:
Inclusion Criteria

* BMI 18 - 28 kg/m2
* SBP 90-140
* DBP 50-90

Exclusion Criteria

* Seizures,
* Orthostatic hypotension

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2010-07; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
AUC0-t, AUC, Cmax, tmax, t1/2, λz, CL/F, Vz/F, MRT (mean residence time) for SLV337 (Part 1 and Part 2) | Part 1: 5 days Part 2: 8 days
AUC0-t, AUC, Cmax, tmax, t1/2, λz, CL/F, Vz/F, MRT (mean residence time) for SLV337 acyl-glucoronide (Part 2) | Part 2: 8 days
Excretion balance of total 14C-radioactivity (Part 2) | Part 2: 8 days
Total 14C-radioactivity (Part 2) | Part 2: 8 days
Metabolic profiling and identification of 14C-labeled parent compound and metabolites of SLV337 in plasma, urine and feces (Part 2) | Part 2: 8 days

SECONDARY OUTCOMES:
Safety and tolerability assessments including adverse events, clinical laboratory tests, ECG and vital signs (Part 1 and Part 2) | Part 1: 19 days Part 2: 15 days

CONTACTS AND LOCATIONS:
Overall Officials: Anita Vanderlaan, Study Director — Abbott Healthcare Products BV
Locations (1):
- Site Reference ID/Investigator# 61345, Zuidlaren, Netherlands